CLINICAL TRIAL: NCT00544960
Title: A Phase 2, Randomized, 2-Arm, Double-Blind Study of AT-101 in Combination With Docetaxel Versus Docetaxel Plus Placebo in Patients With Relapsed or Refractory Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Randomized Phase 2 Study of AT-101 in Combination With Docetaxel in Relapsed/Refractory Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascenta Therapeutics (Industry)
Responsible Party: Brian Wood, Associate Director, Clinical Development, Ascenta Therapeutics
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT-101-CS-204
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: AT101; AT-101; cancer; lung; non-small cell; docetaxel; bcl
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — gossypol acetic acid; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AT-101 and docetaxel
  Interventions: Drug: AT-101 and docetaxel
- 2 (Placebo Comparator): placebo and docetaxel
  Interventions: Drug: placebo and docetaxel

INTERVENTIONS:
Drug: AT-101 and docetaxel — AT-101 30 mg bid on days 1, 2, and 3 of each 21 day cycle, docetaxel, 75 mg/m2 on day 1 of each 21 day cycle; until progression or unacceptable toxicity develops
  Arms: 1
Drug: placebo and docetaxel — placebo 3 tabs bid on days 1, 2, and 3 of each 21 day cycle, docetaxel, 75 mg/m2 on day 1 of each 21 day cycle; until progression or unacceptable toxicity develops
  Arms: 2

SUMMARY:
This is a double- blind, multicenter, randomized Phase II study to evaluate the efficacy and safety of AT-101 in combination with docetaxel in relapsed/refractory non-small cell lung cancer

DETAILED DESCRIPTION:
Further Study Details provided by Ascenta.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Stage IIIb with pleural/pericardial effusion or Stage IV non-small cell lung cancer (NSCLC).
* Progression of disease after one prior systemic chemotherapeutic regimen for locally advanced or metastatic NSCLC. (Systemic therapies given in the adjuvant setting are counted only if the patient relapses within 6 months of the last cycle of therapy.) In addition to the one prior chemotherapeutic regimen, patients may have received erlotinib in any setting.
* All patients must have measurable disease.
* No unstable or progressive brain metastases.
* Patients may have received prior radiation therapy but they must have recovered from all treatment-related toxicities.
* ECOG performance status 0-1
* Adequate hematologic function
* Adequate liver and renal function
* Ability to swallow oral medication

Exclusion Criteria:

* Prior chemotherapy regimen containing docetaxel.
* Active secondary malignancy.
* Uncontrolled concurrent illness including, but not limited to: serious uncontrolled infection, symptomatic congestive heart failure (CHF), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements.
* Failure to recover from toxicities related to prior therapy (e.g., surgery, radiation, chemotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
duration of disease remission | 12 months

SECONDARY OUTCOMES:
number of participants with adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, MD, Study Chair — Ascenta Therapeutics, Inc.
Locations (18):
- Research Site, Durham, North Carolina, United States
- Russia (10):
  - Research Site, Arkhangelsk
  - Research Site, Chelyabinsk
  - Research Site, Kaliningrad
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Sites (4), Saint Petersburg
  - Research Site, Samara
  - Research Site, Stavropol
  - Research Site, Voronezh
  - Research Site, Yekaterinburg
- Ukraine (7):
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Luhansk
  - Research Site, Uzhhorod
  - Research Site, Zaporizhzhya